CLINICAL TRIAL: NCT03859882
Title: Polymorphisms and Efficiency of Caffeine on Performances During Total Sleep Deprivation un Healthy Subject. Multicentric, Versus Placebo, Randomised, Cross Over, Double Blind Study
Brief Title: Protocol PERCAF 2018
Acronym: PERCAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol PERCAF 2018
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Sleep; Caffeine; Polymorphism
Keywords: sleep deprivation; cognition; attention
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): Caffeine 5 mg/kg/day in 2 administration (08:00 and 14:00) per day
  Interventions: Other: Sleep deprivation
- placebo (Placebo Comparator): in 2 administration (08:00 and 14:00) per day
  Interventions: Other: Sleep deprivation

INTERVENTIONS:
Other: Sleep deprivation — 40 hours of continuous awaking in the sleep laboratory in order to compare before and after sleep deprivation for each treatment (Caffeine vs. placebo).

SUMMARY:
In this multicentric controlled study, we aims to evaluate effect of caffeine on mental performances during a sleep deprivation protocol. Genetic polymorphisms are considered as a covariable.

DETAILED DESCRIPTION:
Coffee is the most consumed arousing substance in the world. Caffeine is used as a natural countermeasure to maintain the performance of sleep deprived subjects. However, the effectiveness of caffeine is characterized by a large individual variability, also observed on side effects. This variability could notably be related to polymorphisms of the adenosine receptor 2a gene (ADORA2A) and Tumor Necrosis Factor-alpha, a pro-inflammatory cytokine whose increase is observed during sleep deprivation.

This study, under conditions of total sleep deprivation in the laboratory (40 hours of continuous awakening), examine the cross-influence of two polymorphisms (ADORA2A: rs5751876 and TNF-alpha: rs1800629) on the sensitivity to caffeine and on the degradation of attentional performances. Physical performance, mental performance, immuno-inflammatory responses and the occurrence indesirable effects will be evaluate.

This work aims to understand the mechanisms that contribute to increasing individual vulnerability and promoting protective countermeasures. The purpose of this project is to improve the recommendations concerning the daily use of caffeine and during periods of prolonged awakening, particularly in the military environment.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject

Exclusion Criteria:

* Treatment
* History of cardiovascular, psychiatric, pneumologic, haematologic, cancerology disease
* Nonvoluntary
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Psychomotor vigilance test Speed | Change from Baseline Psychomotor vigilance test Speed at day 2 after 24 hours awaking
  Speed at the Psychomotor vigilance test test

SECONDARY OUTCOMES:
Cognitive performance | Change from Baseline at day 2 after 25 hours awaking
  Number of errors at executive performance test
Force -velocity | Change from Baseline at day 2 after 32 hours awaking
  Power at the force-velocity test

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut de recherche biomedical des armées, Brétigny-sur-Orge
  - Hotel Dieu, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Lorgeril B, Tardo-Dino PE, Bourrilhon C, Quiquempoix M, Drogou C, Mateo L, Erblang M, Colin P, Van Beers P, Chennaoui M, Gomez-Merino D, Sauvet F. Impact of acute caffeine intake on local tolerance to cold before and after total sleep deprivation. Exp Physiol. 2025 Sep;110(9):1254-1270. doi: 10.1113/EP092356. Epub 2025 Mar 27. PMID 40150834
- [Derived] Pauchon B, Beauchamps V, Gomez-Merino D, Erblang M, Drogou C, Beers PV, Guillard M, Quiquempoix M, Leger D, Chennaoui M, Sauvet F. Caffeine Intake Alters Recovery Sleep after Sleep Deprivation. Nutrients. 2024 Oct 11;16(20):3442. doi: 10.3390/nu16203442. PMID 39458438
- [Derived] Drogou C, Sauvet F, Erblang M, Leger D, Thomas C, Chennaoui M, Gomez-Merino D; Investigators group. Effects of Acute Caffeine Intake on Insulin-Like Growth Factor-1 Responses to Total Sleep Deprivation: Interactions with COMT Polymorphism - A Randomized, Crossover Study. Lifestyle Genom. 2023;16(1):113-123. doi: 10.1159/000529897. Epub 2023 Jun 6. PMID 37279709
- [Derived] Erblang M, Drogou C, Gomez-Merino D, Rabat A, Guillard M, Beers PV, Quiquempoix M, Boland A, Deleuze JF, Olaso R, Derbois C, Prost M, Dorey R, Leger D, Thomas C, Chennaoui M, Sauvet F. Genetics and Cognitive Vulnerability to Sleep Deprivation in Healthy Subjects: Interaction of ADORA2A, TNF-alpha and COMT Polymorphisms. Life (Basel). 2021 Oct 19;11(10):1110. doi: 10.3390/life11101110. PMID 34685481
- [Derived] Erblang M, Sauvet F, Drogou C, Quiquempoix M, Van Beers P, Guillard M, Rabat A, Trignol A, Bourrilhon C, Erkel MC, Leger D, Thomas C, Gomez-Merino D, Chennaoui M. Genetic Determinants of Neurobehavioral Responses to Caffeine Administration during Sleep Deprivation: A Randomized, Cross Over Study (NCT03859882). Genes (Basel). 2021 Apr 10;12(4):555. doi: 10.3390/genes12040555. PMID 33920292